CLINICAL TRIAL: NCT03465150
Title: Creation of a Monocentric Cohort of Patients Treated for Acne at the Nantes University Hospital: the COPACNE Cohort.
Brief Title: Creation of a Monocentric Cohort of Patients Treated for Acne at the Nantes University Hospital
Acronym: COPACNE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0218
Record Dates: First submitted 2018-02-05; First posted 2018-03-14 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Acne
Keywords: Acne; Cohort; prospective; risk factors
MeSH Terms: conditions — Acne Vulgaris | interventions — Acne RA-1,2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: acne — Patient with acne
  Other Names: acne vulgaris

SUMMARY:
With 24 million results associated with Google's searchon keywords "severe acne", Pr Dreno's team understand better thatthis disease, which affects many French people, is a real concern of Public Health and not a "forced evil" of the adolescent period, which will eventually resolve itself. Acne does not affect the vital prognosis, but its psychosocial impact is major and should not be underestimated. Paradoxically, despite the high prevalence of acne, few quality epidemiological studies have been published. Physicians are often helpless when faced with patients' questions. They often need a lot of explanations, especially on the factors aggravating this dermatosis, which greatly affects their quality of life.

This cohort, the first of its kind in France, will determine the predictive factors of therapeutic response, endogenous and environmental factors impacting on the severity of acne assess the quality of life and psychological impact of acne patients, determine the patient's course of care and the associated costs. Pr Dreno's team will also build up a bio collection (bacteriological samples).

DETAILED DESCRIPTION:
All patients going for the first time in specialized consultation "acne" at Nantes University Hospital , and who meet the inclusion criteria will be included in the COPACNE cohort. Inclusion will take place at the first consultation, after information and agreement of the patient and, if applicable, his or her legal representatives. The frequency of each patient's follow-up visits will be determined on a case-by-case basis according to the patient's medical needs (generally, the interval between 2 visits is between 1 and 4 months).

ELIGIBILITY:
Inclusion Criteria:

* Patient with acne
* Patient (or parents/guardians for minors) who are not opposed to participating in the cohort.
* Subjects affiliated to an appropriate health insurance

Exclusion Criteria:

* Dermatosis of the face other than acne
* Refusal to participate by the minor or parent/guardian
* Adults under a legal protection regime (guardianship, trusteeship, judicial safeguard)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients going for the first time in specialized consultation "acne"
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2033-02-28 (Estimated); Study Completion 2033-12-28 (Estimated)

PRIMARY OUTCOMES:
Measure of Acne stage | 2 years
  composite criteria. the scale is GEA for Global Evaluation Acne Scale with 0 no acne to 5 severe acne

SECONDARY OUTCOMES:
assessing patients' quality of life | 2 years
  composite criteria. CADI score is calculated by summing the score of each question resulting in a possible maximum of 15 and a minimum of 0. The higher the score, the more the quality of life is impaired.
cost of acne illness | 2 years
  reimbursement data relating to hospitalizations and care in town recorded by the Health Insurance in the SNIIRAM database.
Bacteriological sample to find Propionibacterium acnes, Hormonal check-up on blood sample | 2 years
  Correlation between bacterial and blood samples and the efficacity of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte DRENO, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France